CLINICAL TRIAL: NCT06221189
Title: An Acceptance and Commitment Therapy - Caregiver Support Program (ACT-CSP) for Family Caregivers of Patients Receiving Palliative Care: A Feasibility Study
Brief Title: ACT-CSP for Family Caregivers of Palliative Care Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The end of the funding to the project on 30 April 2024.
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shatin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ACT PC Caregivers
Record Dates: First submitted 2023-11-29; First posted 2024-01-24 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2023-11

CONDITIONS: Caregiver Burden
Keywords: Palliative Care; Caregiving; Acceptance and Commitment Therapy
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-CSP (Experimental): Three sessions of acceptance and commitment therapy.
  Interventions: Behavioral: ACT-CSP
- Usual Care (No Intervention): Usual treatment provided at the participating site.

INTERVENTIONS:
Behavioral: ACT-CSP — The ACT treatment will consist of three 45 to 60-min weekly sessions to be delivered to the caregiver in an individual format via online videoconferencing application e.g. ZOOM or WhatsApp within 3 weeks. The ACT-CSP can be delivered via face-to-face on request. Each session has a specific content with pre-planned materials and mindfulness exercises and metaphors. Psychological-based homework will be assigned at the end of each session. The components of ACT process will be emphasized in the intervention programme, which include perspective taking, self-as-context and defusion (i.e. recognizing worry thoughts as thoughts only), identifying values and acceptance of present-moment experience with respect to the values, and committed action.
  Arms: ACT-CSP

SUMMARY:
The goal of the study is to test the feasibility, acceptability and preliminary efficacy of an acceptance and commitment therapy for supporting caregiver programme (ACT-CSP) on reduction of caregiver burden, anxiety and depressive symptoms and enhancement of caregiving self-efficacy, resilience and quality of life by ACT when compared to usual care, for caregivers of palliative care patients.

DETAILED DESCRIPTION:
This study will employ a pilot randomized controlled trial recruiting caregivers of palliative care patients to receive either a 3-week acceptance and commitment therapy for supporting caregiver programme (ACT-CSP) plus usual care (n = 15) or usual care only (n = 15). The components of acceptance and commitment therapy process will be emphasized in the intervention programme, which include perspective taking, self-as-context and defusion (i.e. recognizing worry thoughts as thoughts only), identifying values and acceptance of present-moment experience with respect to the values, and committed action. The ACT-CSP will be delivered by a trained ACT facilitator. Participants will be followed up at Week 6 and Week 8 after recruitment to collect data for assessing the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18;
* Self- or patient-identified as a family caregiver of an adult patient receiving palliative care at the study site
* Have been taking care of the patient in the past 3 months;
* Able to communicate in Cantonese at the time of recruitment;
* Have access to internet and videoconferencing device such as mobile phone;
* Have caregiver burden as measured by Caregiver Strain Index (CSI) ≥ 7.

Exclusion Criteria:

* Mentally incompetent (Mini-Mental State Examination (MMSE) < 23),
* Participating in regular psychosocial interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Chinese version of the 13-item Caregiver Strain Index | Baseline, Week 6 and Week 8
  Items are rated on a yes (1) or no (0) response, with the total score ranges from 0-13 and higher scores indicating higher caregiver burden

SECONDARY OUTCOMES:
The Patient Health Questionnaire-4 (PHQ-4) | Baseline, Week 6 and Week 8
  The scale scores range from 0 to 12, with higher scores indicating higher levels of anxiety and depression.
The Chinese version of the 18-item modified Caregiver Inventory | Baseline, Week 6 and Week 8
  The scale covers 3 dimensions: Care of the Care Recipient (7 items), Managing information and Self-care (7 items), and Managing emotional interaction with care recipient (4 items). The first two dimensions have scores ranging from 7 to 63 while the last dimension has scores ranging from 4 to 36, with higher scores indicating higher levels of self-efficacy in that dimension.
The 10-item Chinese version of the Connor-Davidson Resilience Scale | Baseline, Week 6 and Week 8
  The overall scores range 0-40, with higher scores indicating higher levels of resilience
The 10-item version of the Singapore caregiver quality of life | Baseline, Week 6 and Week 8
  The overall scores range 0-40, with higher scores indicating higher levels of quality of life

OTHER OUTCOMES:
The 15-item Brief Experiential Avoidance Questionnaire | Baseline, Week and Week 8
  The overall scores range 15-90, with higher scores indicating lower levels of psychological flexibility
Satisfaction to the treatment received | Week 6
  One item on a 0-10 VAS scale, with higher scores indicating higher levels of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Doris YP Leung, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not readily shared because permission to use the data by other researchers has to seek approval from the ethical committee. Requests to access IPD should be directed to PI for further consideration and seeking approval from ethical committee.